CLINICAL TRIAL: NCT06766227
Title: Developing a Smoking Cessation Mobile App. in Arabic: A Pilot Randomized Trial for Efficacy.
Brief Title: Smoking Cessation App. in Arabic
Acronym: iEndSmokin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yarmouk University (Other)
Responsible Party: Principal Investigator, Ola Ali Soudah, Assistant Professor, Yarmouk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-2023
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Smoking Cessation
Keywords: mHealth, Smoking, Cigarette, Behavioral intervention, low-middle income countries
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Experimental): The smoking cessation app will be downloaded and explained to all intervention arm participants after a 2-week run-in period and baseline assessment completion. The smoking cessation app will help smokers set a plan, know how to stop either immediately or progressively, monitor their smoking status and progression, give them tips to overcome cravings, prevent relapses, and aid their mood changes during the cessation trial. The app will provide electronic content, tips, and exercises in written or video-recorded forms. All app content will be evidence-based; based on clinical guidelines and interventions proven in medical literature to be effective. Clinical guidelines used are the "Treating Tobacco Use and Dependence ("2008 update"), and the WHO guidelines. Psychological exercises will be based on CBT which has been shown to reduce smoking rate.
  Interventions: Behavioral: iEndSmokin App
- Education Group (Active Comparator): Three sessions will be provided to the control group one each week for the first month of the study. The first session will take place after a 2-week run-in period following the randomization. All sessions will take place at the Yarmouk University campus or virtually via Zoom in Arabic by a trained research assistant for smoking cessation counseling. The sessions will be educational sessions about smoking health risks, why you should stop, how to stop, and skills and strategies for dealing with withdrawal symptoms.
  Interventions: Behavioral: Educational Session

INTERVENTIONS:
Behavioral: iEndSmokin App — Mobile Health App that includes educational material and psychological programs based on CBT.
  Arms: App Group
Behavioral: Educational Session — It will include lectures and distribution of educational material about smoking health risks and strategies to quit.
  Arms: Education Group

SUMMARY:
Smoking remains a significant global health challenge, causing over 8 million deaths annually, with the burden predominantly in low- and middle-income countries. Jordan experiences some of the highest smoking rates worldwide, contributing to substantial health risks and premature mortality. Despite the prevalence of mobile health (mHealth) applications for smoking cessation, few have supported the Arabic language and none have been evaluated for their efficacy. Our main goal is to develop a culture-sensitive mHealth app in Arabic for smoking cessation and test its efficacy.

DETAILED DESCRIPTION:
Jordan's smoking rates remain among the highest globally despite various initiatives such as smoke-free policies, advertising bans, increased tobacco taxes, and health promotion programs. Mobile health (mHealth) apps have proven effective in delivering education, monitoring health, supporting diagnoses, and acting as therapeutic platforms, overcoming barriers like location, scheduling, and cost. In Jordan, 90% of the population owns smartphones. High-quality apps typically include features like education, goal-setting, progress tracking, skill-building exercises, and community support. Smoking cessation apps' success rates reached up to 27%, where abstinence rates range from 11% to 40.9% within six months.

Treatment guidelines for smoking cessation and/or Psychological therapeutic models such as cognitive behavior therapy (CBT), acceptance commitment therapy (ACT), and mindfulness were infrequently or partially addressed in most Apps. CBT-based smoking-cessation apps are suggested to be more effective. However, adherence to evidence-based guidelines in these apps is low including most commercially available apps. Long-term studies to evaluate App effectiveness and sustainability are scarce. Smoking cessation Apps studies from low-middle-income countries had poor quality, including small sample size, weak designs, and methodological problems, and can't be generalizable across different geographic areas. There is a limited number of smoking cessation Apps in Arabic with no studies testing their efficacy. The Arabic language is widespread, there are about 360.2 people Arabic is their native language encompassing 22 countries. Therefore, the smoking cessation App in Arabic shows an exciting promise for lowering smoking rates at a low cost and convenient setting and thereby preventing tobacco-related premature deaths.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be students attending Yarmouk University recruited through emails and flyers distributed to all offer the University's Faculties. Participation will be on a voluntary base. Only students who fulfill the following criteria will be invited to participate in the study. The inclusion criteria are: 1) a Yarmouk University student, 2) aged 18 years old and above, 3) smoked ≥5 cigarettes a day for the past year (25), 4) have a smartphone (iOS or Android), and 4) express willingness to quit smoking.

Exclusion Criteria:

* The exclusion criteria are: 1) non-Arabic speaker, 2) have certain conditions that interfere with the intervention like blindness or deafness, 3) have clinical depression or mental illness, 4) smoke only hookah, or 5) participate in another smoking cessation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Successful quit attempt | 3 months
  A successful smoking quit event is defined as follows: Participants reported 30 days' abstinence from smoking and all nicotine/tobacco products (Hookah, e-cigarettes, HEETS, cigars, gums …etc.), and very low level of nicotine level (account for second-hand smoking levels) will be considered translated into 30-point abstinence prevalence, and the normal nicotine level in saliva or blood level. Smoking status was the self-reported response to the question "When was the last time you smoked or even tried a cigarette?" Responses choices were "Earlier today", "24 hours ago", "2-7 days ago", "8-30 days ago", and "Over 30 days ago". Salivary or blood Cotinine level test is sensitive to nicotine level for 48-72 hrs. and the samples can be stored for up to three months without jeopardizing the validity of the test

SECONDARY OUTCOMES:
Reduction in Smoking Rate | 3 months
  7-day point prevalence abstinence outcome or decrease in daily cigarettes use

CONTACTS AND LOCATIONS:
Locations (1):
- Yarmouk University, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soudah O, Aldalal'ah M, Alsabbah A, Khasawneh H, Khayyat O, Klaib AF, Alrefai S, Megdadi M. Developing and testing a smoking cessation app in Arabic language: A pilot randomized trial study protocol. Digit Health. 2025 Sep 12;11:20552076251378436. doi: 10.1177/20552076251378436. eCollection 2025 Jan-Dec. PMID 40949668